CLINICAL TRIAL: NCT07336472
Title: A Phase I/II, Multicenter, Open-label Study of IBI3003 in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of IBI3003 in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fortvita Biologics (USA)Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3003A101
Record Dates: First submitted 2026-01-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IBI3003 (Experimental): Participants will receive IBI3003 treatment until death, disease progression, intolerable toxicity, start of a new anticancer treatment, withdrawal of consent for study participation, or end of the study or for a maximum of 24 months, whichever occurs first.
  Interventions: Drug: IBI3003

INTERVENTIONS:
Drug: IBI3003 — Participants will receive IBI3003 treatment until death, disease progression, intolerable toxicity, start of a new anticancer treatment, withdrawal of consent for study participation, or end of the study or for a maximum of 24 months, whichever occurs first.

SUMMARY:
This is a phase 1/2 multicenter, open-label, first-in-human study of IBI3003. It includes a phase 1 dose escalation and expansion section to identify maximum tolerated dose(MTD)/recommended Phase 2 Dose(RP2D) of IBI3003, plans to enroll 54~360 subjects, and a phase 2 stage to explore efficacy, safety and tolerability of IBI3003 at RP2D in multiple myeloma

ELIGIBILITY:
Inclusion Criteria

Participants in Parts 1 & 2 must satisfy all of the following criteria to be enrolled in the study:

1. Age ≥18 years.
2. Documented initial diagnosis of multiple myeloma according to IMWG diagnostic criteria.

   Multiple myeloma is defined as clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma, and any one or more of the following myelomadefining events:
   * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically: Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or corrected serum calcium >2.75 mmol/L (>11 mg/dL) Renal insufficiency: creatinine clearance <40 mL/min or serum creatinine >177 μmol/L (>2 mg/dL) Anemia: hemoglobin value of >2 g/dL below the lower limit of normal, or a hemoglobin value <10 g/dL Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT
   * Any one or more of the following biomarkers of malignancy:

   Clonal bone marrow plasma cell percentage ≥60% Involved: uninvolved serum free light chain ratio ≥100 (involved FLC level must be

   ≥100 mg/L) >1 focal lesions on MRI studies (at least 5 mm in size)
3. Relapsed or refractory measurable multiple myeloma (R/R MM) following prior treatment with ≥3 lines of systemic anti-myeloma therapy that include at least a proteasome inhibitor (PI), an immunomodulatory drug (IMiD) agent, and an anti-CD38-based therapy, and with limited or no therapeutic options that are likely to offer a favorable risk/benefit profile; participants must be relapsed or refractory to their last anti-myeloma regimen.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
5. At least one of the following measurable disease indicators:

   * Serum M-protein ≥5 g/L (for IgA and IgD subtypes, quantitative immunoglobin measurements could be used as substitutions for M-protein)
   * Urine M-protein ≥200 mg/24h
   * Serum free light chain (FLC) test: affected FLC level ≥100 mg/L and abnormal serum FLC ratio (<0.26 or >1.65)
6. Adequate hematologic, hepatic, renal and cardiac function:

   * Blood count: absolute neutrophil count ≥1.0×10^9/L, hemoglobin ≥70 g/L, and platelet count ≥50×10^9/L (values must be achieved without growth factors or blood transfusions within 7 days prior to first dose)
   * Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both ≤2.5× upper limit of normal (ULN) and total bilirubin (TBIL) ≤1.5×ULN
   * Renal function: calculated creatinine ≥30 mL/min by the Cockcroft-Gault Equation
   * Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%
7. Life expectancy ≥3 months.
8. Women of childbearing potential and fertile men who are sexually active must agree to use a highly effective method of contraception (<1% / year failure rate) during the study and for 90 days after the last dose level of study drug. Contraception must be consistent with local regulations or standards regarding the use of birth control methods by participants participating in clinical trials. Women and men must agree not to donate or bank eggs (ova, oocytes) or sperm, respectively, during the study and for 90 days after the last dose level of study drug.
9. Participants with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.
10. Willing and able to adhere to the complete schedule of assessments and all prohibitions and restrictions specified in this protocol

Exclusion Criteria

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
2. Active amyloidosis, plasma cell leukemia, Waldenstrom macroglobulinemia, POEMS syndrome, or solitary plasmacytoma, or smoldering multiple myeloma (MM) as defined by the IMWG criteria.
3. Spinal cord compression that results in limited self-care at present or within 6 months prior to informed consent, or that is expected to cause such limitations during Study participation.
4. History of primary immunodeficiency.
5. Current or previous other malignancy within 3 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
6. Allogeneic hematopoietic stem cell transplantation within the last 6 months, or autologous stem cell transplantation within the last 3 months prior to the first administration of the study drug.
7. History of organ transplantation.
8. Active graft-versus-host disease.
9. Thromboembolism or cerebrovascular events (e.g., myocardial infarction, unstable angina, transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with complications of central venous access], or pulmonary embolism) within 6 months prior to the first dose of study drug.
10. Pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation.
11. Known allergies, hypersensitivity, or intolerance to IBI3003 or its excipients (refer to Investigator's Brochure).
12. Prior toxicities that have not resolved to ≤Grade 1 prior to study treatment administration except for stable chronic toxicities (≤Grade 2) not expected to resolve (e.g., stable Grade 2 peripheral neurotoxicity)
13. Prior antitumor therapy as follows, prior to the first dose of study drug:

    * Gene modified adoptive cell therapy (e.g., chimeric antigen receptor modified T cells, natural killer cells) within 8 weeks.
    * Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 14 days or at least 5 half-lives, whichever is longer.
    * Antibody treatment (e.g., monoclonal antibody, bispecific antibody) for multiple myeloma within 21 days.
    * Cytotoxic therapy (including antibody-drug conjugates) within 14 days.
    * Proteasome inhibitor therapy within 14 days Immunomodulatory agent therapy within 7 days.
    * Radiotherapy within 21 days. However, if the radiation field covered ≤5% of the bone marrow reserve, the participant is eligible irrespective of the end date of radiotherapy.
    * Cancer vaccine received within 3 months.
14. Use of immunosuppressive therapy within 28 days of the start date of study treatment.

    Immunosuppressive therapy includes, but is not limited to, cyclosporine A, tacrolimus, and mycophenolate mofetil, but does not include corticosteroids given as part of an antimyeloma regimen. Participants receiving corticosteroids must be at a dose level ≤10 mg/day of prednisone equivalent for at least 7 days prior to the start of study treatment administration.
15. Live or live attenuated vaccine administered within 4 weeks prior to start of study treatment, or anticipated need for live or live attenuated vaccine during the study.
16. Uncontrolled diseases, including:

    * Uncontrolled infection or infection requiring systemic antibiotics, antivirals or antifungals within one week prior to first administration of the study drug;
    * Known human immunodeficiency virus (HIV) infection, or HIV positive (HIV 1/2 Ab positive);
    * For participants in mainland China, acute or chronic active hepatitis B (HBsAg positive and/or HBcAb positive with HBV DNA titer ≥104 copies/mL or ≥2000 IU/mL) or C (HCV Ab positive with HCV RNA>103 copies/mL). For participants outside of mainland China, active, latent or incompletely treated infection with HBV or HCV;
    * Failed to complete anti-tuberculosis therapy at any point prior to C1D1; active tuberculosis infection, or still on anti-tuberculosis therapy;
    * Active syphilis infection requiring treatment;
    * Symptomatic congestive heart failure Grade II-IV (New York Heart Association [NYHA]), symptomatic or uncontrolled arrhythmias, QTc interval (calculate using the Fridericia formula) >480 ms, or personal or family history of congenital long/short QT syndrome;
    * Uncontrollable hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg);
    * Active autoimmune diseases, including but not limited to inflammatory bowel disease, autoimmune hepatitis, demyelinating lesions, extensive dermatitis, immunerelated interstitial pneumonia, or Grave's disease requiring antithyroid medication control (vitiligo, or hypothyroidism requiring hormone replacement therapy, type I diabetes requiring only insulin replacement therapy and no other systemic therapy in the past 2 years are eligible); Presence of clinically uncontrolled pleural/peritoneal effusions (participants who do not require regular drainage or who do not demonstrate significant re-accumulation of effusion for at least 72 hours after the most recent drainage can enroll).
17. Major surgery within 2 weeks prior to the first dose of study treatment, not fully recovered from any prior surgery, or has non-minor surgery anticipated during the time the participant is expected to receive study drug or within 2 weeks after the last dose of study drug administration.
18. Participating in any other interventional clinical research except an observational (noninterventional) study or the survival follow-up phase of an interventional study.
19. Currently pregnant or breastfeeding.
20. Any condition that would, in the Investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
21. Inability to comprehend or unwilling to sign the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 30 days post last dose
  Number of patients who Experienced related AEs from the first dose until 30 days after the last dose
Dose limiting toxicities (DLTs) | Up to 28 days post first dose
  To evaluate the safety and tolerability of IBI3003
ORR | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
To determine the maximum tolerated dose (MTD) and the recommended Phase 2 Dose (RP2D) of IBI3003 | up to 24 months
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 Dose (RP2D) of IBI3003

SECONDARY OUTCOMES:
Incidence and characterization of anti-drug antibody (ADA). | up to 24 months
  To evaluate the immunogenicity of IBI3003
Preliminary efficacy including objective response rate (ORR) | up to 24 months
  objective response rate. To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
To evaluate minimal residual disease (MRD) negativity rates. MRD negativity rate. | up to 24 months
  To evaluate minimal residual disease (MRD) negativity rates.
efficacy estimates sCRR | up to 24 months
  stringent complete response rate. To evaluate other efficacy estimates of IBI3003 in the participant population.
Incidence of TEAEs | up to 24 months
  To evaluate the safety of IBI3003 in the participant population.
half-life (T1/2) | up to 24 months
  To characterize the pharmacokinetic (PK) profile of IBI3003.
time to maximum concentration (Tmax) | up to 24 months
  time to peak concentration. To characterize the pharmacokinetic (PK) profile of IBI3003.
maximum concentration (Cmax) | peak plasma concentration. To characterize the pharmacokinetic (PK) profile of IBI3003.
  up to 24 months
area under the curve (AUC) | up to 24 months
  area under the curve. To characterize the pharmacokinetic (PK) profile of IBI3003.
complete response rate (CRR) | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
very good partial response rate (VGPRR) | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
duration of response (DoR) | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
disease control rate (DCR) | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
time to response (TTR) | To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
  up to 24 months
progression free survival (PFS). | up to 24 months
  To evaluate the preliminary efficacy of IBI3003 in the specified participant population.
SAEs | up to 24 months
  serious adverse events (SAEs) Adverse events will be assessed by investigator(s) To evaluate the safety of IBI3003 in the participant population.
changes in laboratory parameters | up to 24 months
  To evaluate the safety of IBI3003 in the participant population.
physical examination findings | up to 24 months
  A complete physical examination will include: general appearance, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose, and pharynx), lymph nodes, thyroid, musculoskeletal (including spine and extremities), genital/anal, and neurological assessments, if indicated. Clinically significant abnormal findings at screening will be recorded as medical history or AE based on the investigator's analysis and judgment.To evaluate the safety of IBI3003 in the participant population.
vital signs | up to 24 months
  Collection of vital signs will include temperature in ℃, measurement tool is physiological parameter.To evaluate the safety of IBI3003 in the participant population.